CLINICAL TRIAL: NCT00312312
Title: Does Specific Immunotherapy Possess Immunomodulative Effects at the Bronchial Mucosa Level Among Adults With Atopic Diseases?
Brief Title: Allergy Towards Grass and Bronchial Inflammation - Related to Immunotherapy and Exhaled Nitrogen Oxide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SITNO
Record Dates: First submitted 2006-04-05; First posted 2006-04-10 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2006-09

CONDITIONS: Asthma, Bronchial; Allergic Rhinitis; Hypersensitivity, Immediate
Keywords: Asthma; Allergic rhinitis; Atopy; Exhaled nitric oxide; Specific immunotherapy; Atopic diseases
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Hypersensitivity, Immediate

INTERVENTIONS:
Biological: Specific immunotherapy

SUMMARY:
The purpose of this study is to evaluate the immunomodulatory effect of treatment of allergic rhinitis symptoms with specific immunotherapy by measurement of pulmonary inflammatory markers, and among others, exhaled nitric oxide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old
* Skin prick test or RAS test and physical examination conclude that the patient will have a beneficial effect from specific immunotherapy

Exclusion Criteria:

* Other diseases except atopic disease
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-03; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Skin prick test
Spirometry
Methacholine provocation of the pulmonary system
Exhaled nitric oxide
Immunoglobulin E (IgE) status
Sputum examination
Condensation of exhaled air

SECONDARY OUTCOMES:
Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, M.D., M.D.Sci, Principal Investigator — Lungeforskningsenheden v/Bispebjerg hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark